CLINICAL TRIAL: NCT06641752
Title: Evaluation of the Accuracy of Capillary Versus Venous CO Measurement in Subjects With Suspected Carbon Monoxide Poisoning: a Prospective, Multicenter, Diagnostic, Controlled Study.
Brief Title: Evaluation of CO Intoxication Rate, by CAPillary HbCO
Acronym: COCAP
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC24_0511; 2024-A02162-45 (Other: ANSM (IDRCB))
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Carbon Monoxide Intoxication
Keywords: Intoxication; Carbon monoxyde; Carboxyhemoglobin; COHb; Carboxyhemoglobin capillary
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: The study population must correspond to the research inclusion criteria:
  Adult patient admitted to the emergency department, presenting with one or more clinical signs (asthenia, headache, nausea, vomiting, loss of consciousness, etc.) and a history compatible with CO intoxication (collective symptoms, notion of smoke, activation of a detector, etc.)
  Interventions: Diagnostic Test: Blood drop sampling

INTERVENTIONS:
Diagnostic Test: Blood drop sampling — The process: blood drop sampling Technique: capillary sampling Frequency: Once Time: 5 minutes Sample collection volume: 1mL Total collection volume: 1 mL

SUMMARY:
The main goal of COCAP is to compare COHb (carboxyhemoglobin) levels measured from venous or arterial samples with those measured from capillary samples in patients suspected of Carbon Monoxide intoxication.Patient participation in the study will be limited to capillary sampling (approx. 5-15 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted to emergency department
* Presenting one or more clinical signs (asthenia, headache, nausea, vomiting, loss of consciousness, etc.) and a history compatible with CO intoxication (collective symptoms, notion of smoke, activation of a detector, etc.).

Exclusion Criteria:

* Minors
* Patients under protective supervision (safeguard of justice, curatorship, guardianship)
* Incarcerated patients
* Pregnant or breast-feeding women
* Patients refusing to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients admitted to adult emergency departments with suspected carbon monoxide intoxication.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Determine the accuracy of capillary HbCO measurement (compared with venous or arterial HbCO) in patients with suspected CO poisoning. | 15 minutes
  The main goal will be determined by the mean bias and limits of agreement between capillary and venous (or arterial) sampling (Bland-Altman analysis).

SECONDARY OUTCOMES:
Determine the diagnostic performance of capillary measurement | 15 minutes
  Determine the sensitivity, specificity, ROC curve, area under the ROC curve, positive and negative predictive values and likelihood ratios (positive and negative) of capillary measurement for the diagnosis of CO intoxication. The linear correlation coefficient between venous (or arterial) HbCO and capillary HbCO will also be calculated.
Assess the technical difficulties of different blood sampling processes (Measurement of the number of attempts and failure rate for samples) | 15 minutes
Assess the technical difficulties of different blood sampling processes (Measurement of the time required to take each sample) | 15 minutes
Analyse the technical difficulties associated with the analysis of the two samples (Time between sampling and HbCO result) | 15 minutes
Analyse the technical difficulties associated with the analysis of the two samples (percentage of samples that cannot be analysed by the laboratory) | 15 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU d'Angers, Angers, Loire-Atlantique
  - Nantes University Hospital, Nantes, Loire-Atlantique

IPD SHARING:
Plan to Share IPD: Undecided